CLINICAL TRIAL: NCT01895439
Title: Phase II Study: Use of Autologus Mesenchymal Stem Cells in Multiple Sclerosis Patients Who do Not Respond to Conventional Treatment
Brief Title: Safety and Efficacy Study of Autologus Bone Marrow Mesenchymal Stem Cells in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Fatima Jamali, Researcher, University of Jordan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSUJCTC
Record Dates: First submitted 2013-06-24; First posted 2013-07-10 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Bone marrow derived Mesenchymal Stem Cells; Multiple Sclerosis; Oligodendrocytes; Neuroimmunology; Autoimmune disease
MeSH Terms: conditions — Multiple Sclerosis; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSCs injection (Experimental): Autologous bone marrow derived stem cells injected intrathecally to enrolled MS patients
  Interventions: Biological: Autologous Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells

SUMMARY:
1. Expanding and priming Bone Marrow (BM)- Mesenchymal Stem Cells (MSCs) to a clinical scale according to Good Laboratory Practice using xenogenic free media instead of the previously used FCS.
2. Assessing the safety of injecting autologous BM-MSCs to Multiple Sclerosis (MS)patients who fail to respond to conventional treatment.
3. Assessing the therapeutic benefits on the participants in the trial as per established methods.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of definite MS according to the revised McDonald Criteria.
* Expanded Disability Status Scale (EDSS) ≤ 6
* Failure of standard medical therapy
* Disease duration of at least three years prior to enrollment.

Exclusion Criteria:

* Pregnant and lactating women
* Previous treatment with immunosuppressive agents in the last 12 months prior to enrollment
* Recent MS relapse in the month prior to enrollment
* Treatment with oral or parenteral steroids for any cause in the month prior to enrollment
* Significant systemic medical disorders including cardiac, renal, hepatic, hematologic, immunologic or endocrine disorders
* Previous treatment with interferons or glatiramer acetate in the 3 months prior to enrollment
* Any contra-indication for magnetic resonance imaging (MRI) or gadolinium contrast.
* Positive serology for HIV, Hepatitis B or Hepatitis C
* Any history of malignancy or exposure to radiation at any time prior to enrollment
* Any contra-indication to lumbar puncture
* Severe cognitive impairment that would interfere with the patient's ability to understand and sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The number of patients with any relevant side effects observed | 18 months
  Assessing the safety of autologous Mesenchymal Stem Cells injection

SECONDARY OUTCOMES:
Assessing the therapeutic benefits of the injected Autologous Mesenchymal Stem Cells by Magnetic Resonance Imaging (MRI) and ophthalmological tests. | 18 months
  For every patient tests would be performed at baseline and repeated at 3, 6, and 18 months post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD., Study Director — Cell Therapy Center; Said Dahbour, MD., Principal Investigator — Jordan University Hospital
Locations (1):
- Cell Therapy Center, Jordan University Hospital, Amman, Jordan